CLINICAL TRIAL: NCT04506099
Title: Transcutaneous Intercostal Nerve Stimulation in Spinal Cord Injury
Acronym: TINS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of study staff
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Spinal Cord Injury Medicine Research Director, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-20-0048
Record Dates: First submitted 2020-07-16; First posted 2020-08-10 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Neuropathic Pain; SCI - Spinal Cord Injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized sham-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study participants will be blinded to the stimulation parameters of the TINS. The research assistant/investigator will apply the electrodes and the PI will be blinded the stimulation setting as well. Unblinding is expected to occur after the 2 month follow up, at which point both subject and PI will be made aware of their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TINS Active (Active Comparator): Electrical stimulation will be applied to the T6-T11 levels of intercostal nerves, as close to the level directly below the level of injury as possible. For example, a T7 level of injury will have TINS applied to the T8 level. A T2 level of injury will have TINS applied to the T6 level. Electrodes 2 inch by 4 inch will be placed according to anatomic landmarks with the negative electrode applied to the lateral ribcage and the positive electrode applied to the ventral aspect, verified with contraction of the rectus abdominis. The intensity level will be set to the amperage immediately under the threshold for motor contraction. If there is no contraction seen, patients will be excluded. In addition, if the patient perceives pain, the intensity will be lowered until comfortable. Stimulation frequency of 20 Hz and pulse width of 200ms in continuous mode will be used.
  Interventions: Device: TINS Active protocol
- Sham protocol (Sham Comparator): Electrical stimulation will be applied to the T6-T11 levels of intercostal nerves, as close to the level directly below the level of injury as possible until contraction is seen in the rectus abdominis. Stimulation frequency of 20 Hz and pulse width of 200ms in continuous mode will be used. Electrodes 2 inch by 4 inch will be placed according to anatomic landmarks with the negative electrode applied to the lateral ribcage and the positive electrode applied to the ventral aspect. The intensity level will be set to 1mA . If there is no contraction seen, patients will be excluded. In addition, if the patient perceives pain, the intensity will be lowered until comfortable.
  Interventions: Device: Sham protocol

INTERVENTIONS:
Device: TINS Active protocol — Electrical stimulation will be applied to the T6-T11 levels of intercostal nerves, as close to the level directly below the level of injury as possible. Electrodes 2 inch by 4 inch will be placed according to anatomic landmarks with the negative electrode applied to the lateral ribcage and the positive electrode applied to the ventral aspect, verified with contraction of the rectus abdominis. The intensity level will be set to the amperage immediately under the threshold for motor contraction. If there is no contraction seen, patients will be excluded. In addition, if the patient perceives pain, the intensity will be lowered until comfortable. Stimulation frequency of 20 Hz and pulse width of 200ms in continuous mode will be used.
  Arms: TINS Active
Device: Sham protocol — Electrical stimulation will be applied to the T6-T11 levels of intercostal nerves, as close to the level directly below the level of injury as possible until contraction is seen in the rectus abdominis. Stimulation frequency of 20 Hz and pulse width of 200ms in continuous mode will be used. Electrodes 2 inch by 4 inch will be placed according to anatomic landmarks with the negative electrode applied to the lateral ribcage and the positive electrode applied to the ventral aspect. The intensity level will be set to 1mA . If there is no contraction seen, patients will be excluded. In addition, if the patient perceives pain, the intensity will be lowered until comfortable.
  Arms: Sham protocol

SUMMARY:
The purpose of this study is to determine the safety, feasibility, and effectiveness of electric stimulation of the nerves along the intercostal nerves on pain and spasticity in spinal cord injury patients.

DETAILED DESCRIPTION:
Neuromodulation techniques are safely used as a treatment for neuropathic pain in chronic SCI. Neuromodulation techniques have also been safely and successfully used to strengthen the abdomen in stroke patients.10 Most similar to our TINS protocol is transcutaneous tibial nerve stimulation (TTNS), which has shown to mitigate the development of neurogenic bladder in acute SCI.6 However, neuromodulation is rarely performed in acute SCI, and, to our knowledge, neuromodulation has not been performed to prevent the development of chronic neuropathic pain. There has been little published regarding the effects of electric stimulation upon the trunk in acute SCI as a prevention for chronic neuropathic pain and spasticity. Gaps in the knowledge which we intend to fill are:

1. Safety and feasibility of TINS in acute SCI during inpatient rehabilitation.
2. Effectiveness of a 2-week TINS protocol in acute SCI based on changes between admission, discharge, and weekly numerical pain scores and spasticity questionnaire scores in those with TINS compared to sham TINS for 2-months.
3. Analysis of neuropathic pain medication dosages in those with and without TINS at admission, discharge, and 2 months post-discharge, and evaluation of morbidity at 2- months post-discharge

ELIGIBILITY:
Inclusion Criteria:

* Acute tSCI paraplegia within 4 weeks of injury (n=22)
* 18-75 years old
* Neurologic levels T1-T10
* English speaking
* Admitted to TIRR with pain medications
* TINS can elicit visible or palpable abdominal muscle contraction

Exclusion Criteria:

* Subjects with pacemakers, defibrillators, insulin pumps, and similar devices
* History of peripheral neuropathy
* History of premorbid symptoms of peripheral neuropathy (numbness and/or tingling in the lower extremities, sharp/jabbing/burning pain in the lower extremities, sensitivity to touch, lack of coordination, lack of sensation, muscle weakness, etc.)
* History of nervous system disorder (i.e. prior SCI, stroke, brain injury, degenerative diseases such as Parkinson's disease, etc.)
* Ventilator dependent respiration
* Inability to speak
* Non-English speakers
* Pregnancy
* History of chronic pain
* Intolerant to electric stimulation
* Intolerant to the trial sessions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with morbidity as measured by infections | Admission
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking infections
Number of participants with morbidity as measured by infections | 4-weeks post injury
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking infections.
Number of participants with morbidity as measured by infections | 2-month follow-up
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking infections.
Number of participants with morbidity as measured by burns. | Admission
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking burns.
Number of participants with morbidity as measured by burns. | 4-weeks post injury
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking burns.
Number of participants with morbidity as measured by burns. | 2-month follow-up
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking burns.
Number of participants with morbidity as measured by urgent transfers. | Admission
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking urgent transfers
Number of participants with morbidity as measured by urgent transfers. | 4-weeks post injury
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking urgent transfers
Number of participants with morbidity as measured by urgent transfers. | 2-month follow up
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking urgent transfers
Number of participants with morbidity as measured by spasticity scores per usual care. | Admission
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking spasticity scores recorded per usual care
Number of participants with morbidity as measured by spasticity scores per usual care. | 4-weeks post injury
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking spasticity scores recorded per usual care
Number of participants with morbidity as measured by spasticity scores per usual care. | 2-month follow-up
  Observe the safety of using TINS during acute inpatient rehabilitation by prospectively tracking spasticity scores recorded per usual care

SECONDARY OUTCOMES:
Number of participants with improved spasiticy scores as measured by PENN SPASM FREQUENCY SCALE (PSFS) | Baseline
  Contains clinically relevant core questions concerning SCI-related pain. This is a 2 component self-report measure of the frequency of reported muscle spasms which is commonly used to quantify spasticity. Developed to augment clinical ratings of spasticity and provide a more comprehensive understanding of an individual's spasticity status. The first component is a 5 point scale assessing the frequency with which spasms occur ranging from "0 = No spasms" to "4 = Spontaneous spasms occurring more than ten times per hour". The second component is a 3 point scale assessing the severity of spasms ranging from "1 = Mild" to "3 = Severe". The second component is not answered if the person indicates they have no spasms in part. Lower scores indicate better outcomes.
Number of participants with improved spasiticy scores as measured by PENN SPASM FREQUENCY SCALE (PSFS) | 2-month follow-up
  Contains clinically relevant core questions concerning SCI-related pain. This is a 2 component self-report measure of the frequency of reported muscle spasms which is commonly used to quantify spasticity. Developed to augment clinical ratings of spasticity and provide a more comprehensive understanding of an individual's spasticity status. The first component is a 5 point scale assessing the frequency with which spasms occur ranging from "0 = No spasms" to "4 = Spontaneous spasms occurring more than ten times per hour". The second component is a 3 point scale assessing the severity of spasms ranging from "1 = Mild" to "3 = Severe". The second component is not answered if the person indicates they have no spasms in part. Lower scores indicate better outcomes.
Number of participants with decreased pain medication dosage compared at discharge and 2-month follow-up. | 4-weeks post injury
  Compare number of participants with decreased pain medication dosage at discharge and 2-month follow-up.
Number of participants with decreased pain medication dosage compared at discharge and 2-month follow-up. | 2-month follow-up
  Compare number of participants with decreased pain medication dosage at discharge and 2-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, Principal Investigator — UTHealth
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackery A, Tator C, Krassioukov A. A global perspective on spinal cord injury epidemiology. J Neurotrauma. 2004 Oct;21(10):1355-70. doi: 10.1089/neu.2004.21.1355. PMID 15672627
- [Background] McNeill DL, Carlton SM, Hulsebosch CE. Intraspinal sprouting of calcitonin gene-related peptide containing primary afferents after deafferentation in the rat. Exp Neurol. 1991 Dec;114(3):321-9. doi: 10.1016/0014-4886(91)90158-9. PMID 1748206
- [Background] McNeill DL, Hulsebosch CE. Intraspinal sprouting of rat primary afferents after deafferentation. Neurosci Lett. 1987 Oct 16;81(1-2):57-62. doi: 10.1016/0304-3940(87)90340-5. PMID 3696474
- [Background] Diamond J, Foerster A. Recovery of sensory function in skin deprived of its innervation by lesion of the peripheral nerve. Exp Neurol. 1992 Jan;115(1):100-3. doi: 10.1016/0014-4886(92)90229-j. No abstract available. PMID 1728554
- [Background] Gwak YS, Hulsebosch CE. Neuronal hyperexcitability: a substrate for central neuropathic pain after spinal cord injury. Curr Pain Headache Rep. 2011 Jun;15(3):215-22. doi: 10.1007/s11916-011-0186-2. PMID 21387163
- [Background] Stampas A, Korupolu R, Zhu L, Smith CP, Gustafson K. Safety, Feasibility, and Efficacy of Transcutaneous Tibial Nerve Stimulation in Acute Spinal Cord Injury Neurogenic Bladder: A Randomized Control Pilot Trial. Neuromodulation. 2019 Aug;22(6):716-722. doi: 10.1111/ner.12855. Epub 2018 Oct 3. PMID 30284350
- [Background] Hatch MN, Cushing TR, Carlson GD, Chang EY. Neuropathic pain and SCI: Identification and treatment strategies in the 21st century. J Neurol Sci. 2018 Jan 15;384:75-83. doi: 10.1016/j.jns.2017.11.018. Epub 2017 Nov 16. PMID 29249383
- [Background] Ataoglu E, Tiftik T, Kara M, Tunc H, Ersoz M, Akkus S. Effects of chronic pain on quality of life and depression in patients with spinal cord injury. Spinal Cord. 2013 Jan;51(1):23-6. doi: 10.1038/sc.2012.51. Epub 2012 May 1. PMID 22547044
- [Background] Johnson MI, Bjordal JM. Transcutaneous electrical nerve stimulation for the management of painful conditions: focus on neuropathic pain. Expert Rev Neurother. 2011 May;11(5):735-53. doi: 10.1586/ern.11.48. PMID 21539490
- [Background] Ko EJ, Chun MH, Kim DY, Yi JH, Kim W, Hong J. The Additive Effects of Core Muscle Strengthening and Trunk NMES on Trunk Balance in Stroke Patients. Ann Rehabil Med. 2016 Feb;40(1):142-51. doi: 10.5535/arm.2016.40.1.142. Epub 2016 Feb 26. PMID 26949681
- [Background] Nichols ME, Meador KJ, Loring DW, Poon LW, Clayton GM, Martin P. Age-related changes in the neurologic examination of healthy sexagenarians, octogenarians, and centenarians. J Geriatr Psychiatry Neurol. 1994 Jan-Mar;7(1):1-7. doi: 10.1177/089198879400700101. PMID 8192823
- [Background] https://www.nscisc.uab.edu/Public/Facts%202015.pdf
- [Background] Dubeau CE. The aging lower urinary tract. J Urol. 2006 Mar;175(3 Pt 2):S11-5. doi: 10.1016/S0022-5347(05)00311-3. PMID 16458733
- [Background] http://www.emsci.org/index.php/project/the-project/time-schedule
- [Background] Chartier-Kastler EJ, Denys P, Chancellor MB, Haertig A, Bussel B, Richard F. Urodynamic monitoring during percutaneous sacral nerve neurostimulation in patients with neurogenic detrusor hyperreflexia. Neurourol Urodyn. 2001;20(1):61-71. doi: 10.1002/1520-6777(2001)20:13.0.co;2-d. PMID 11135383
- [Background] Bellucci CH, Wollner J, Gregorini F, Birnbock D, Kozomara M, Mehnert U, Schubert M, Kessler TM. Acute spinal cord injury--do ambulatory patients need urodynamic investigations? J Urol. 2013 Apr;189(4):1369-73. doi: 10.1016/j.juro.2012.10.013. Epub 2012 Oct 12. PMID 23069382
- [Background] Buchele G, Och B, Bolte G, Weiland SK. Single vs. double data entry. Epidemiology. 2005 Jan;16(1):130-1. doi: 10.1097/01.ede.0000147166.24478.f4. No abstract available. PMID 15613958
- [Background] Verrills P, Vivian D, Mitchell B, Barnard A. Peripheral nerve field stimulation for chronic pain: 100 cases and review of the literature. Pain Med. 2011 Sep;12(9):1395-405. doi: 10.1111/j.1526-4637.2011.01201.x. Epub 2011 Aug 3. PMID 21812906
- [Background] Petersen EA, Slavin KV. Peripheral nerve/field stimulation for chronic pain. Neurosurg Clin N Am. 2014 Oct;25(4):789-97. doi: 10.1016/j.nec.2014.07.003. Epub 2014 Aug 15. PMID 25240665